CLINICAL TRIAL: NCT00551772
Title: An Open-Label, Randomised, Two-Part Crossover Study to Assess the Pharmacokinetics of a Single Dose of SB-742457 Formulated as a Capsule and a Tablet in Healthy Elderly Volunteers.
Brief Title: A Study To Assess The Pharmacokinetics Of SB-742457 Formulated As A Capsule And A Tablet In Healthy Elderly Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AZ3110291
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2008-12-25 (Estimated); Status verified 2008-12

CONDITIONS: Alzheimer's Disease
Keywords: Bio-availability, healthy elderly volunteers
MeSH Terms: conditions — Alzheimer Disease | interventions — 3-benzenesulfonyl-8-piperazin-1-ylquinoline

INTERVENTIONS:
Drug: SB-742457

SUMMARY:
SB-742457 is a 5HT6 receptor antagonist that is in development for the symptomatic treatment of mild to moderate Alzheimer's disease . To date, all clinical trials have been conducted using a capsule formulation of SB-742457. However, it is intended to conduct all futures studies with a tablet formulation. The aim of this study is to assess the pharmacokinetic profile of SB-742457 and its major metabolites following single doses of both the capsule and tablet formulations.

ELIGIBILITY:
Inclusion criteria:

* Men or surgically sterile or post-menopausal women
* Healthy as judged by a responsible physician. No clinically significant abnormality identified on the medical or lab evaluation.
* BMI between 18.5 and 32.0 kg/m2

Exclusion criteria:

* A positive pre-study urine screen for drugs of abuse
* Abuse of alcohol
* Subjects who smoke more than 10 cigarettes or equivalent a day.
* Use of prescription drugs as well as herbal and dietary supplements within 7 days prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Where participation in the study would result in donation of blood in excess of 500ml within a 56 day period.
* Has a history or presence of gastro-intestinal, hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* The subject has received an investigational drug or participated in another research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Known or suspected history of seizures, including febrile seizures, unexplained recent loss of consciousness or history of significant head trauma with loss of consciousness.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-08

PRIMARY OUTCOMES:
To characterise pharmacokinetics ( AUC(0-inf) and Cmax ) of SB-742457 from pre-dose to 96 hours following single doses formulated as a capsule and a tablet. | pre-dose to 96 hours

SECONDARY OUTCOMES:
To assess safety and tolerability (adverse events, blood pressure, heart rate, 12-lead ECG, blood haematology/clinical chemistry and urinalysis) of SB-742457 following single doses formulated as a capsule and a tablet over the 6 week study period. | 6 week study period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, PhD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Evansville, Indiana, United States